CLINICAL TRIAL: NCT03550482
Title: ONCOXIN® and Quality of Life in Cancer Patients in a Real World Setting Study
Brief Title: Oncoxin® and Quality of Life in Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-5
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-05

CONDITIONS: Gastric Cancer Stage II; Non-small Cell Lung Cancer Stage II; Non-small Cell Lung Cancer Stage III; Gastric Cancer Stage III
Keywords: Oncoxin; Nutritional supplement; Chemotherapy; Oxidative stress; Antioxidant
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Study multicenter open-label nonrandomized clinical trial in two parallel groups with a 20-day treatment period. No follow-up period was intended. Following visits were scheduled: Visit 1 - the first day of 2nd and further course of ACT before ACT drugs administration; Visit 2 - 7±1 days before next course of ACT; Visit 3 - the day of next course of ACT before ACT drugs administration (21±3 days after Visit 1).
  It is expected, that the proportion of patients with MCID improvement in total SDS ESAS was 50% in ONCX group and 20% in control group (with baseline total SDS ESAS of 30 points). Based on patients' allocation as 2:1 in comparison groups for the ONCX and control groups, respectively, alpha 0.05 and power not less than 0.9 data of 120 patients has to be analyzed. With the dropout of 25% 150 patients has to be included in the study (100 ONCX/50 controls).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oncoxin® (Experimental)
  Interventions: Dietary Supplement: ONCOXIN®
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: ONCOXIN® — Adjuvant chemotherapy regimen (XELOX or paclitaxel+carboplatin) + Oncoxin 25 ml twice daily for 20 days. In case of nausea/vomiting after ONCX use patients were advised to dilute it in water, juice or milk. Patients with BMI <20 and serum albumin levels <30 g/l received nutritional support.
  Arms: Oncoxin®

SUMMARY:
It is expected that additional support with certain micronutrients may improve prognosis, decrease the frequency of side effects and complications and maintain high relative dose intensity of anticancer treatments. Food supplement ONCOXIN (ONCX) contains amino acids, vitamins, minerals and biologically active substances of natural origin with high immunostimulatory and antioxidant activity. Present study is a real world experience study intended to evaluate the efficacy of ONCX in cancer patients.

DETAILED DESCRIPTION:
The study was conducted at 9 centers across the Russia and Kazakhstan. Patients were allocated in 2:1 comparison groups for the ONCX and control groups, respectively. A total of 133 patients were enrolled in the study; 84 in the ONCX group and 49 as controls.

ONCX contains microelements, vitamins, amino acids and certain naturally occurring, biologically active substances.

It is expected that additional support with certain micronutrients may improve prognosis, decrease the frequency of side effects and complications and maintain the Quality of life in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients who had signed an informed consent.
2. Males and females aged 50-70 y/o
3. Gastric cancer IIB-IIIC, Non-small cell lung cancer IIB-IIIA
4. R0 surgery
5. Adjuvant chemotherapy (ACT) required, 2nd and further course of ACT, XELOX regimen of ACT for gastric cancer and paclitaxel+carboplatin regimen for non-small cell lung cancer.
6. Body mass index (BMI) ≥ 15, serum albumin ≥ 25 g/l.
7. Eastern Cooperative Oncology Group performance status ≤ 2

Exclusion Criteria:

1. Severe concomitant diseases or conditions that may complicate or make impossible the patient's participation in the study, or make it difficult to interpret the clinical data (including mental disorders, severe infectious and parasitic diseases and intolerability to any of the ONCX components).
2. The patient's family or official relations with a member of staff of the study center.
3. The patient's failure to assess his/her physical and/or emotional condition.
4. The patient's failure to comply with the study requirements.
5. The patient's refusal to participate in the study and pregnancy or lactation.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Quality of life improvement | 20 days
  The proportion of patients who had an improvement in the QoL corresponding to the minimal clinically important difference (MCID) that any patient was able to feel at Visits 2 in total SDS ESAS (6 points within patient change for improvement)

SECONDARY OUTCOMES:
Emotional Quality of life | 20 days
  emotional SDS ESAS domains
Toxicity produced by Chemotherapy | 20 days
  Common toxicity criteria NCI-CTC. Common Terminology Criteria for Adverse Events (AE) is a descriptive terminology which can be utilized for Adverse Event reporting. A grading (severity) scale is provided for each AE term.
Toxicity produced by Chemotherapy | 20 days
  Body Mass Index (BMI) combined with albumin. High body mass index (BMI) has been inconsistently associated with overall survival. Preoperative body mass index, blood albumin and triglycerides predict survival for patients with gastric cancer.
Physical Quality of Life | 20 days
  Physical SDS ESAS scores
Nutritional level | 20 days
  Serum albumin level measures

CONTACTS AND LOCATIONS:
Locations (9):
- Kazakhstan (2):
  - Kazakh Research Institute of Oncology and Radiology, Almaty
  - State Municipal Enterprise on the Right of Economic Management "Almaty Oncology Center" of Almaty Healthcare Administration, Almaty
- Russia (7):
  - State-funded Institution of Khanty-Mansiysk Regional Clinical Hospital, Ugra, Tyumen Oblast
  - Medical Center "EVIMED" LLC, Chelyabinsk
  - State-funded Healthcare Institution Oncologic Clinical Dispensary No.1, Moscow
  - The Loginov Moscow Clinical Scientific Center, www.mknc.ru, Moscow
  - Medical University "Reaviz", Samara
  - Non-government Healthcare Institution " Hospital of JSC Russian Railways Hospital at the Station Smolensk, Smolensk
  - State-funded Institution "Surgut Regional Hospital", Surgut

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Kaidarova DR, Kopp MV, Pokrovsky VS, Dzhugashvili M, Akimzhanova ZM, Abdrakhmanov RZ, Babich EN, Bilan EV, Byakhov AV, Gurov SN, Koroleva IA, Mochalova AS, Povaga SS, Raigorodsky MV, Saifullin AS, Sanz E, Petrovskiy FI. Multicomponent nutritional supplement Oncoxin and its influence on quality of life and therapy toxicity in patients receiving adjuvant chemotherapy. Oncol Lett. 2019 Nov;18(5):5644-5652. doi: 10.3892/ol.2019.10868. Epub 2019 Sep 13. PMID 31641390